CLINICAL TRIAL: NCT05956652
Title: Observational Study on the Efficacy and Safety of Transcatheter Implantation of Hydra Biological Aortic Prosthesis
Brief Title: Hydra Registry - Italy Experience
Status: Recruiting | Type: Observational
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: Clinica Di Montevergine (Other)
Responsible Party: Sponsor
Other Study IDs: Hydra-IT, V1.0, 02/03/2022
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; TAVI; Hydra
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Hydra Transcatheter Aortic Valve System — The Hydra device is self-expanding transcatheter aortic valve consists of a self-expanding nitinol frame and three bovine pericardial leaflets in supra-annular position.

SUMMARY:
Hydra-IT is a multicenter observational study aim to collect clinical, procedural and follow-up data and evaluate the short, medium and long term results of Hydra TAVI System in patient with severe aortic stenosis.

DETAILED DESCRIPTION:
Hydra-IT is a multicenter observational study conducted across different centres in Italy. The primary objective of the study is to evaluate the safety and efficacy of transcatheter aortic valve implantation and clinical outcome in patients treated with Hydra device. Secondary objective is to evaluate the long term (up to 5 years) effectiveness and the quality of treatment using Hydra device. Patients with severe stenosis symptomatic of the native aortic valve or bioprosthesis in a degenerated aortic position will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe symptomatic native aortic valve stenosis and candidates for the TAVI procedure based on the evaluation of the Heart Team
* Ability to understand and provide informed consent for inclusion in the study

Exclusion Criteria:

* Contraindication to TAVI: e.g. evidence of intracardiac mass, thrombus or vegetation, endocarditis.
* Refusal by the patient to participate in the study
* High probability of non-adherence to required follow-ups

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with severe aortic valve stenosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | 30 days

SECONDARY OUTCOMES:
All-cause mortality | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Cardiovascular mortality, valve-related mortality, and non-cardiovascular mortality
All stroke | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Disabling and non-disabling stroke
Disabling stroke | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Myocardial infarction | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Life-threatening or disabling bleeding | 30 days
Major vascular complications | 30 days
Acute kidney injury (Stage 2 or 3) | 30 days
New permanent pacemaker implantation (PPM) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Paravalvular Leak (PVL) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Effective Orifice Area (EOA) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Mean aortic valve gradient | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
New York Heart Association (NYHA) functional classification | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Angelo Cioppa, Principal Investigator — Montevergine Clinic, Mercogliano, Italy
Locations (4):
- Italy (4):
  - Fondazione Poliambulanza Istituto, Brescia
  - Montevergine Clinic, Mercogliano, Italy, Mercogliano
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan
  - Università degli studi di Padova, Padua

IPD SHARING:
Plan to Share IPD: No